CLINICAL TRIAL: NCT00804232
Title: Childhood Diabetes - Family Based Health Interventions for Child Health
Brief Title: Childhood Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Collaborators: Lund University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: principal investigators: inger Hallsgtröm; Gun Forsander, Inger Hallstrom, Lund University; Gun Forsander, Sahlgrenska University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DiabetesVardal
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes, Type I
Keywords: Diabetes type1; children
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): effects on child health of family-based home care compared to traditional hospital-based care,
  Interventions: Behavioral: childhood diabetes
- 2 (Experimental): effects on child health of family-based psychological treatment compared to traditional hospital-based treatment
  Interventions: Behavioral: childhood diabetes

INTERVENTIONS:
Behavioral: childhood diabetes — the intervention compares three different regimes for children newly diagnosed with type 1 diabetes: (1) traditional hospital based care, (2) intensive psychological support to the family, and (3) home based family psychosocial support. A further aim is to identify families were the child runs the risk of decreased metabolic control and to give those families increased support.

SUMMARY:
Purpose of the study:

To compare three different regimes for children newly diagnosed with type 1 diabetes: (1) traditional hospital based care, (2) intensive psychological support to the family, and (3) home based family psychosocial support. A further aim is to identify families were the child runs the risk of decreased metabolic control and to give those families increased support.

Specific objectives:

The main objectives of the study are:

1. to analyse the effects on child health of family-based home care compared to traditional hospital-based care, and
2. to analyse the effects on child health of family-based psychological treatment compared to traditional hospital-based treatment.

The main focus will be on child health and changes in child health. Several variables will be collected for these purpose (see instruments, below), the main variable being the child's metabolic control. We will also analyse effects on the amount and content of (1) parental efforts (absenteeism from work; time use which is conditional on the child's diabetes etc), and (2) formal health care utilisation of the home-based care and psychological treatment, respectively, compared to traditional care.

DETAILED DESCRIPTION:
Purpose of the study:

To compare three different regimes for children newly diagnosed with type 1 diabetes: (1) traditional hospital based care, (2) intensive psychological support to the family, and (3) home based family psychosocial support. A further aim is to identify families were the child runs the risk of decreased metabolic control and to give those families increased support.

Specific objectives:

The main objectives of the study are:

(3) to analyse the effects on child health of family-based home care compared to traditional hospital-based care, and (4) to analyse the effects on child health of family-based psychological treatment compared to traditional hospital-based treatment.

The main focus will be on child health and changes in child health. Several variables will be collected for these purpose (see instruments, below), the main variable being the child's metabolic control. We will also analyse effects on the amount and content of (1) parental efforts (absenteeism from work; time use which is conditional on the child's diabetes etc), and (2) formal health care utilisation of the home-based care and psychological treatment, respectively, compared to traditional care.

Methods:

Design:

The study is planned to include four parts: one historical control group including data for metabolic control from the Swedish diabetes register for children (SWEDIABKIDS), two randomised controlled trials at two different university hospitals in Sweden (Lund and Gothenburg), and one prospective control group at one region hospitals (Helsingborg). Data will be collected at inclusion and after six, 12 and 24 months after diagnosis. We plan a longitudinal follow-up five and ten year after diagnosis concerning metabolic control and complications.

Inclusion criteria: children, aged 3 - 15, newly diagnosed with diabetes mellitus; no other chronic illnesses; Swedish as mother tongue; no siblings with type 1 diabetes; not objects for social interventions.

Analysis:

The main analysis is that of the differences in child health (main variable: HbA1c) between intervention and control groups. Analysis of variance (ANOVA) will be applied.

Instruments and data:

Metabolic control:

P-glucos (self-monitoring) during the first two years. Weekly random chosen twenty-four hour graph. HbA1c monthly during the first two years. From this a yearly mean HbA1c is established.

Reports according to SWEDIABKIDS/NDRBarn: for example weight, length, BMI, insulin (time, dose, type), blood pressure, U-albumin, severe hypoglucaemia, and cetoacidosis, number of hospitalisations.

Background variables:

Age, civil status, number of persons in the family, education, occupation, level of employment.

Quality of life, well-being, and health:

PedsQL Generic Core Scales, Child self-report (Adolescent 13-18 years, Child 8-12 years), Young Child, Parent proxy report (5-7 years) (Varni & PedsMetrics/The PedsQL™)..

PedsQL, Diabetes module (Varni & PedsMetrics/The PedsQL™). Children 8-18 years, parents proxy report (children 5-7 years).

SF 36, Health Utility Index. Satisfaction with care PedsQL, Health Care Satisfaction Generic Module. Parents. (Varni & PedsMetrics/The PedsQL™).

Family impact and family climate The PedsQLTM Family Impact Module. Parents. Physical, emotional, social and cognitive function, communikation, anxiety, daily activities, and family relations. (Varni & PedsMetrics/The PedsQL™).

Diabetes Family Behavior Scale.

Diabetes Family Conflict:

Family climate. Shows changes from therapeutic interventions (Hansson, 1991). Mastery. (Pearlin, Menaghan, Lieberman & Mullan, 1981). Controll in daily life and the possibility to achive individual goals.

THU-5, (Targeting Hassles and Uplifts- five items, Erlandsson & Eklund, 2003). Parents experiences of hassles and uplifts in daily life.

THU-3 (Targeting Hassles and Uplifts- three items) Costs of social welfare-during and after the initial hospitalisation Hospital costs during hospitalisation. Professionals' time use which is conditional on the child's diabetes for the different regiments.

Number and time for out patient visits/home visits. Number and time for telephone contacts.

Psychosocial Assessment:

Psychosocial Assessment Tool, (The Children's hospital of Philadelphia, Division of Oncology, 2004) meassure psychosocial variables, family interplay, and family function.

Absenteeism from work and school Familjens diabetesrelaterade frånvaro från arbete och skola Parental and child's absenteeism from work and school related to the diabetes. 12 och 24 mån.

ELIGIBILITY:
Inclusion Criteria:

* children, aged 3 - 15
* newly diagnosed with diabetes mellitus
* no other chronic illnesses
* Swedish as mother tongue
* no siblings with type 1 diabetes
* not objects for social interventions

Exclusion Criteria:

-

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: the child's metabolic control as shown in HbA1C | 6 months, 1 year, 2 year, 5 year

SECONDARY OUTCOMES:
Quality of life, Satisfaction with care, Family impact and family climate, psychological variables, parental absenteeism from work; time use which is conditional on the child's diabetes etc), formal health care utilisation | 6 months, 1 year, 2 year, 5 year

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Queen Silvia's Childrens' hospital, Gothenburg
  - Lund University Childrens' hospital, Lund

REFERENCES:
- [Derived] Tiberg I, Lindgren B, Carlsson A, Hallstrom I. Cost-effectiveness and cost-utility analyses of hospital-based home care compared to hospital-based care for children diagnosed with type 1 diabetes; a randomised controlled trial; results after two years' follow-up. BMC Pediatr. 2016 Jul 15;16:94. doi: 10.1186/s12887-016-0632-8. PMID 27421262
- [Derived] Tiberg I, Carlsson A, Hallstrom I. A Methodological Description of a Randomised Controlled Trial Comparing Hospital-Based Care and Hospital-Based Home Care when a Child is Newly Diagnosed with Type 1 Diabetes. Open Nurs J. 2011;5:111-9. doi: 10.2174/18744346011050100111. Epub 2011 Nov 18. PMID 22371819